CLINICAL TRIAL: NCT00584207
Title: Radiofrequency Ablation of Uterine Fibroids
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Unsufficient referrals for recruitment
Sponsor: University of California, Davis (Other)
Responsible Party: John McGahan, M.D., University of California, Davis Dept. of Radiology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200412085
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Uterine Fibroids
Keywords: uterine fibroids
MeSH Terms: conditions — Leiomyoma | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: radiofrequency ablation — Intraoperative RFA of uterine fibroids

SUMMARY:
This research study is being conducted to evaluate the safety and effectiveness of ablation (destruction) of uterine leiomyomas (fibroids) using electrocautery heating guided by ultrasound. We are doing this to look for a less invasive method of treatment for patients with uterine fibroids. One method that is being used in other areas of the body to treat masses is radiofrequency electrocautery. This method may be performed for the treatment of uterine fibroids by placing a small diameter needle through the wall of the vagina into the fibroid guided by an ultrasound probe. An optional approach is to place the needle through the skin of the abdomen into the fibroid guided by an ultrasound probe. Once the needle is in the fibroid, the electrocautery current is applied and the fibroid is destroyed by heating. This would be done before hysterectomy (removal of the uterus). We are trying to test to see if this type of treatment can be applied to uterine fibroids. We are trying to develop radiofrequency electrocautery as one of the methods to treat fibroids without surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosed with uterine leiomyomas (fibroids)
* Patient will undergo surgical hysterectomy
* Patient is willing to sign informed consent form

Exclusion Criteria:

* Patients with acute infection
* Patients with bleeding disorders
* Patients who are not candidates for surgery or general anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-03; Primary Completion 2007-03 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Following the hysterectomy, the study pathologist will perform a histological examination of the treated fibroid specimen to determine the size and volume of the ablation that was created with radiofrequency electrocautery. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: John P. McGahan, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States